CLINICAL TRIAL: NCT01330810
Title: Crossover, Multiple Dose Pharmacokinetics of Two Curcumin Formulations in Healthy Volunteers
Brief Title: Curcumin Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 10-2243
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2011-12

CONDITIONS: Comparative Multidose Pharmacokinetics
Keywords: Pharmacokinetics; Dietary Supplements; Curcumin
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C3 tablet (Active Comparator): 4g C3 tablet
  Interventions: Drug: curcumin
- Meriva (Active Comparator): 2g Meriva powder
  Interventions: Drug: curcumin

INTERVENTIONS:
Drug: curcumin — standardized curcumin supplements containing curcumin, demethoxycurcumin and bisdemethoxycurcumin

SUMMARY:
Each year, there are about 150,000 new colorectal cancer (CRC) cases and 50,000 CRC deaths in the United States. A safe and effective preventive agent could reduce the burden of colorectal cancer as well as reduce the costs associated with screening patients who are at high risk of developing CRC. Preclinical studies strongly suggest that curcumin is active against multiple pathways implicated in tumor initiation, progression, and metastasis. However, little is know how curcumin performs in humans. The investigators propose to enroll 12 healthy volunteers who will undergo blood draw and rectal biopsy after 7 days of curcumin administration. The investigators will look at curcumin preparations with low and high oral bioavailability and calculate the blood and rectal tissue concentrations associated with these two formulations to determine which preparation produces the highest tissue concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years of age
2. BMI 18 - 30 kg/m^2
3. Ability/willing to provide informed consent
4. Good general health

Exclusion Criteria:

1. History of any pancreatic or biliary disease (eg. Familial colorectal cancer syndromes, Ulcerative colitis or Crohn's disease)
2. History of any acute or chronic illness that requires current medical therapy, including active gastrointestinal conditions, that might interfere with drug absorption
3. History of large bowel resection for any reason
4. Diagnosed narcotic or alcohol dependence
5. Women with childbearing potential who do not agree to practice effective birth control.
6. Use of curcumin within the last 14 days
7. Allergy to study agent
8. Individuals with creatinine, AST or ALT above 1.5 times the upper limit of normal at baseline.
9. Personal or inherited bleeding disorders or therapeutic anti-coagulation with warfarin.
10. Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
AUC | 0-48h
  Area under plasma concentration curve from 0-48h using 13 time points.
Cmax | 0-48h
  Maximum curcumin plasma concentration
Tmax | 0-48h
  Time to maximum curcumin plasma concentration
Ke | 0-48h
  Terminal elimination rate
T1/2 | 0-48h
  plasma curcumin concentration half-life
Vd | 0-48h
  Volume of distribution
Test of bioequivalence | 0-48h
  geometric mean ratio of plasma AUC0-48h of the two formulations
bioequivalence of tissue curcumin concentration | 1h
  comparison of curcumin concentration in colorectal tissue at single time point between two formulations

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Asher, MD, MPH, Principal Investigator — UNC
Locations (1):
- UNC Department of Family Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Asher GN, Xie Y, Moaddel R, Sanghvi M, Dossou KS, Kashuba AD, Sandler RS, Hawke RL. Randomized Pharmacokinetic Crossover Study Comparing 2 Curcumin Preparations in Plasma and Rectal Tissue of Healthy Human Volunteers. J Clin Pharmacol. 2017 Feb;57(2):185-193. doi: 10.1002/jcph.806. Epub 2016 Sep 6. PMID 27503249